CLINICAL TRIAL: NCT07167238
Title: An Evaluation of the Effect of Video Game-Based Exercise Training on Functional Exercise Capacity and Respiratory Parameters in Patients With Interstitial Lung Disease
Brief Title: The Effect of Video Game-Based Exercise Training in Patients With Interstitial Lung Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Zeynep Kaçar Akkoç, Principal Investigator, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/353
Record Dates: First submitted 2025-08-15; First posted 2025-09-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial lung disease; Video game; Exercise training; Functional exercise capacity; Respiratory parameters
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Exergaming

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video game-based exercise training (Experimental): In addition to the unsupervised conventional pulmonary rehabilitation program, they will participate in a supervised video game-based exercise protocol twice a week.
  The conventional physiotherapy and rehabilitation program will include posture exercises combined with breathing exercises three times a day, every weekday, and a walking program twice a week, along with breathing exercises. The supervised video game-based exercise program will include five different five-minute breathing labs and breathing games, two days a week, and 40 minutes of Nintendo Wii Fit games, which include lower extremity, upper extremity, and balance exercises.
  Interventions: Behavioral: Virtual reality exercises
- Conventional Pulmonary Rehabilitation (Active Comparator): Only the unsupervised conventional pulmonary rehabilitation (PR) program will be applied on this group. The conventional PR program will include posture exercises combined with breathing exercises three times a day, every weekday, and a walking program twice a week, along with breathing exercises
  Conventional PR program including:
  Breathing exercises (pursed-lip breathing, thoracic expansion, diaphragmatic breathing, breathing control) Postural exercises combined with breathing Walking program (30 min, 2×/week at Borg scale 4-6)
  Interventions: Behavioral: Home exercises

INTERVENTIONS:
Behavioral: Virtual reality exercises — Program Duration: 8 weeks Implementation: The conventional program plus supervised video game-based training sessions.
  Additional Protocol: Video Game-Based Exercises
  1. Breathing Labs - Breathing Games (Slovenia) Frequency: 3 days per week, on non-walking days, supervised at the hospital. Structure: 5 mini-games per session, performed sequentially.
     Exercises:
     Balloon: Weeks 1-4: Level 1; Weeks 5-8: Level 2. Focus on sustained controlled exhalation.
     Plane: Weeks 1-4: ~6 sec breath cycle; Weeks 5-8: ~8 sec breath cycle. Wolf: Weeks 1-4: Easy; Weeks 5-8: Medium. Flowers: Weeks 1-4: Sunflower module; Weeks 5-8: Rose module. Pluto: Weeks 1-4: Easy; Weeks 5-8: Medium. Intensity: Target MBS 4-6/10 for dyspnea and fatigue.
  2. Nintendo Wii / Wii Fit - Functional Training Duration: ~5 minutes per game, 30-40 minutes total per session.
  Games and targets:
  Lower limb/aerobic: Basic Run, Basic Step, Obstacle Course, Island Cycling. Upper limb: Boxing, Canoe. Balance: Rhythm Parade.
  Arms: Video game-based exercise training
Behavioral: Home exercises — Program Duration: 8 weeks Implementation: Home-based, instructed face-to-face at baseline by a physiotherapist, supported with video materials, and monitored with regular feedback.
  A) Posture + Breathing Exercises Frequency: 3 sessions per day (morning, noon, evening)
  Content:
  Shoulder girdle mobilization: Scapular elevation-depression, abduction-adduction (3 sets × 3 repetitions).
  Stretching exercises: Shoulder, cervical, and trunk muscles; 5-second hold at end range.
  Combined with breathing: Inspiration during concentric phase, expiration during eccentric phase.
  B) Breathing Exercises Frequency: 3 sessions per day; 10 repetitions of each exercise per session
  Content:
  Pursed-Lip Breathing, Thoracic Expansion Exercises, Diaphragmatic Breathing, Breathing Control C) Walking Program Frequency: 2 days per week Duration: 30 minutes (5 min warm-up, 20 min walking, 5 min cool-down) Intensity: Self-selected pace targeting Modified Borg Scale (MBS) 4-6/10 for dyspnea.
  Arms: Conventional Pulmonary Rehabilitation

SUMMARY:
The goal of this prospective randomized controlled clinical trial is to evaluate the effects of video game-based physiotherapy and rehabilitation on functional exercise capacity and respiratory parameters in individuals with interstitial lung disease (ILD). The study also aims to compare the outcomes of video game-based rehabilitation with conventional physiotherapy, identify alternative breathing exercises for pulmonary involvement in ILD, and provide scientific evidence to guide clinical practice.

The main questions it aims to answer are:

Does video game-based rehabilitation improve respiratory function parameters in individuals with ILD?

Does video game-based rehabilitation reduce dyspnea and exercise intolerance, thereby improving functional exercise capacity?

Does video game-based rehabilitation increase participation and completion rates in pulmonary rehabilitation programs? Study Design: A total of 42 participants diagnosed with mild-to-moderate ILD will be recruited. Participants will be randomized into two groups (21 in the intervention group, 21 in the control group) using stratified randomization to ensure homogeneity by age, sex, and ILD type.

Arms: 2 (Intervention group and Control group)

Intervention:

Intervention group: Structured video game-based exercise training sessions as part of a pulmonary rehabilitation program.

Control group: Conventional pulmonary rehabilitation program.

Assessments: Respiratory function, functional exercise capacity, and symptom levels will be measured before and after the intervention.

Inclusion criteria:

Diagnosis of mild-to-moderate ILD

Aged 20-70 years

Referral by a treating physician

Willingness and ability to participate

No physical or cognitive barriers to exercise training

Exclusion criteria:

Cardiovascular disease (e.g., acute heart failure, unstable angina, recent myocardial infarction)

Cognitive impairment

History of cerebrovascular event

History of cancer

Withdrawal criteria:

Development of clinical hemodynamic instability

Major surgical complication during the study

Missing ≥ 3 consecutive training sessions in the intervention group

Withdrawal of consent

DETAILED DESCRIPTION:
Interstitial lung diseases (ILDs) are chronic parenchymal disorders characterized by varying degrees of inflammation and fibrosis, leading to exertional dyspnea, exercise intolerance, ventilatory restriction, and reduced health-related quality of life. Beyond pulmonary involvement, patients often experience fatigue, peripheral muscle weakness, anxiety, and reduced participation in daily activities. Pulmonary rehabilitation is a key non-pharmacological strategy for ILD; however, adherence and completion rates remain limited due to barriers such as symptom burden, transportation, and the repetitive nature of conventional exercise training.

Technology-assisted rehabilitation, particularly video game-based training (exergaming), has emerged as a promising strategy to enhance motivation and adherence while preserving the physiological benefits of exercise. Exergaming provides real-time feedback, goal-oriented tasks, and progressive challenges that may improve enjoyment, engagement, and consistency of participation. In respiratory rehabilitation, game-guided breathing exercises may reinforce techniques such as pursed-lip breathing, diaphragmatic breathing, and thoracic expansion, which optimize ventilatory mechanics and potentially reduce dyspnea. Additionally, whole-body functional games can promote aerobic capacity, coordination, and peripheral muscle endurance.

This randomized controlled trial is designed to compare the effects of video game-based rehabilitation combined with conventional physiotherapy versus conventional physiotherapy alone in individuals with mild-to-moderate ILD. A total of 42 participants will be randomized into two parallel arms (intervention and control). The intervention arm will receive supervised video game-based exercise sessions in addition to standard pulmonary rehabilitation, while the control arm will perform conventional home-based physiotherapy and rehabilitation only.

Primary outcomes include changes in respiratory function parameters, functional exercise capacity, and symptom perception before and after the 8-week intervention. The study also aims to examine whether video game-based rehabilitation increases adherence and completion rates compared to conventional programs.

The expected impact of this study is to provide scientific evidence regarding the feasibility, safety, and effectiveness of integrating video game-based rehabilitation into pulmonary rehabilitation for ILD. If successful, this approach may help overcome barriers to participation, improve functional outcomes, and support broader implementation of engaging, patient-centered rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with mild to moderate interstitial lung disease
* Being between the ages of 20 and 70
* Being referred to the study by their physician
* Being willing and able to participate
* Having no physical or cognitive disability that would prevent them from participating in exercise training

Exclusion Criteria:

* Presence of cardiovascular disease (acute heart failure, unstable angina, or recent myocardial infarction, etc.)
* Presence of cognitive impairment that prevents participation in exercise training
* Presence of a history of cerebrovascular accident
* Presence of a history of cancer

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | Day 1 and at the end of the eighth week
  FVC will be measured using a spirometry test. During the assessment, participants will be instructed to take a full breath, and with a nose clip in place, exhale into the spirometer with maximum effort. The procedure will be repeated at least three times, and the best value will be recorded. Results will be expressed in liters (L) and compared to predicted values based on age, height, sex, and ethnicity. A value of ≥80% of the predicted capacity will be considered normal.
Forced Expiratory Volume in 1 Second (FEV₁) | Day 1 and at the end of the eighth week
  FEV₁ is defined as the volume of air that will be exhaled during the first second of a forced expiration after a full inspiration. It will be measured by spirometry and expressed in liters (L). Results will be compared to predicted values calculated according to age, height, sex, and ethnicity. A value of ≥80% of the predicted capacity will be considered normal.
FEV₁/FVC | Day 1 and at the end of the eighth week
  The FEV₁/FVC ratio is defined as the proportion of the forced expiratory volume in the first second (FEV₁) to the forced vital capacity (FVC). It will be measured by spirometry. Results will be expressed as a percentage and compared to predicted values according to age, height, sex, and ethnicity. A value of ≥70% will be considered normal, while lower values will indicate airflow limitation.
Peak Expiratory Flow (PEF) | Day 1 and at the end of the eighth week
  Peak Expiratory Flow (PEF) is defined as the maximum flow rate that will be achieved during a forced expiration after a full inspiration. It will be measured by spirometry and expressed in liters per second (L/s). The procedure will be repeated at least three times, and the best value will be recorded. Results will be compared to predicted values calculated according to age, height, sex, and ethnicity. A value of ≥80% of the predicted capacity will be considered normal.
Lung Diffusion Capacity | Day 1 and at the end of the eighth week
  Diffusing capacity (DLCO) measurement will be performed with the nose closed after the patient has not exercised before the test and has been sitting for at least 5 minutes. Care should be taken to ensure rapid inspiration. Inspiration time should be kept between 2 and 4 seconds. The final expiration should not exceed 4 seconds. Breath-hold times will be measured for all patients as recommended by the European Respiratory Society (ERS) guidelines. Tests with breath-hold times outside the 9-11 second range, inspirations with inspiratory vital capacity (IVC) below 90% during the DLCO maneuver, and measurements with alveolar ventilation below 10% of total lung capacity will be excluded from the study. DLCO measurements will be performed using gas chromatographs, and the results will be recorded as ml/min/mmHg. Hemoglobin-corrected tests will be used as the basis.
Peripheral muscle strength | Day 1 and at the end of the eighth week
  Peripheral muscle strength will be measured using a portable manual muscle strength measurement device (Hoggan MicroFet2 Handheld Dynamometer) for shoulder abductor and adductor, shoulder flexor, extensor, elbow flexor and extensor, hip flexor, extensor, hip abductor, adductor, knee flexor, and extensor muscles. Grip strength will be measured using a handheld dynamometer (Jamar, Nottinghamshire, UK) in a sitting position, with the elbow flexed at 90 degrees and the wrist in neutral. Measurements will be repeated three times for the right and left sides, and the average of the values will be recorded in Newtons (N).
Functional Exercise Capacity | Day 1 and at the end of the eighth week
  Functional exercise capacity will be assessed with the 6-minute walk test (6MWT). Participants are instructed to walk a 30-meter corridor with the goal of covering the longest possible distance in six minutes. Participants are allowed to stop and rest if necessary but are encouraged to continue walking as soon as possible. Participants' heart rate, blood pressure, peripheral oxygen saturation, self-perceived shortness of breath, and lower extremity muscle fatigue are questioned before and after the test. The distance traveled during the six-minute period is recorded. The 6MWT is a valid and reliable test for interstitial lung disease.

SECONDARY OUTCOMES:
Quality of Life score | Day 1 and at the end of the eighth week
  The quality of life score will be assessed using the St. George Respiratory Questionnaire (SGRQ). The SGRQ is a self-assessment questionnaire specific to airway diseases. It consists of 76 questions in three categories. It examines symptoms, activities, and the impact of the disease on daily life. Each section is scored separately from 0 to 100. A score of 0 indicates no impairment in quality of life, while a score of 100 indicates maximum disability and a poor quality of life. So a higher score means a worse outcome.
The Modified Borg Scale Score | Day 1 and at the end of the eighth week
  This scale will be used to evaluate the dyspnea level of the participants. The Modified Borg Scale is scored between 0 and 10. A score of 0 means no shortness of breath at all, while a score of 10 means it's unbearably severe. In other words, a higher score indicates a worse outcome.
Modified Medical Research Council Scale Score | Day 1 and at the end of the eighth week
  This scale will be used to evaluate the dyspnea level of the participants. Modified Medical Research Council Scale (MMRC) is graded from 0 to 4. As the score increases, shortness of breath becomes more severe and functional limitations increase. In other words, a higher score is associated with a worse outcome.
Fatigue status | Day 1 and at the end of the eighth week
  Fatigue status of patients will be evaluated with the Fatigue Severity Scale (FSS). This scale assesses fatigue severity with nine questions. Each question is scored from 1 (completely disagree) to 7 (completely agree). The FSS score is the average of the nine sections. A higher score indicates increased fatigue severity.
Dysfunctional Respiration | Day 1 and at the end of the eighth week
  Dysfunctional respiratory status of patients will be evaluated with the Nijmegen Questionnaire. The Nijmegen Questionnaire is a questionnaire used to identify dysfunctional breathing patterns and unexplained respiratory symptoms. It consists of 16 items scored from 0 to 4. The total score ranges from 0 to 64. A higher total score indicates dysfunctional breathing.
Cognitive Function | Day 1 and at the end of the eighth week
  Patients' cognitive functions will be assessed using the Montreal Cognitive Assessment Scale (MOCA). This scale includes sections assessing executive functions, attention and concentration, memory, language, abstract thinking, visual-spatial skills, orientation, and calculation. The total score is calculated out of 30. The threshold score is 21. Scores of 20 or lower are considered cognitive dysfunction. Higher scores indicate greater cognitive preservation, while lower scores indicate poorer cognitive function.